CLINICAL TRIAL: NCT03622060
Title: A Randomized Comparison of Post-procedural/Pre-hemostasis Intraarterial Nitroglycerin Versus Nicardipine to Reduce Radial Artery Occlusion After Transradial Catheterization
Brief Title: Intraarterial Nitroglycerin Versus Nicardipine and Radial Artery Occlusion
Acronym: NONERAO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hermina Heart Center Kemayoran (Other)
Collaborators: Hermina Hospital Group (Unknown)
Responsible Party: Principal Investigator, Surya Dharma, MD, PhD, NONERAO study, Hermina Heart Center Kemayoran
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HerminaHCK
Record Dates: First submitted 2018-08-01; First posted 2018-08-09 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Radial Artery Injury at Wrist and Hand Level; Occlusion of Artery; Vasodilation
MeSH Terms: conditions — Arterial Occlusive Diseases; Aneurysm | interventions — Nitroglycerin; Nicardipine

STUDY DESIGN:
Intervention Model Description: nitroglycerin and nicardipine
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitroglycerin (Active Comparator): 500 microgram intraarterial Nitroglycerin
  Interventions: Drug: Nitroglycerin
- Nicardipine (Placebo Comparator): 200 microgram intraraterial Nicardipine
  Interventions: Drug: Nitroglycerin

INTERVENTIONS:
Drug: Nitroglycerin — 200 microgram intraarterial nicardipine and 500 microgram nitroglycerin administered before sheath removal
  Other Names: Nicardipine

SUMMARY:
A total of 600 patients undergoing coronary procedures via transradial access using 6F sheath were randomized at the end of the procedure to receive either 250-µg nicardipine or 500-µg nitroglycerin administered to the radial artery through the radial sheath before sheath removal. A continuous patent hemostasis was applied in each patient with the use of an oximetry to maintain an oxygen saturation of >95%, measured in the finger of the accessed arm until compression device was totally removed. The primary outcome is early RAO which was evaluated by color duplex ultrasonography of the accessed arteries at the day after the radial procedure. Secondary outcome was the change of blood pressure at 2-3 minutes after drug administration. Radial artery angiogram was performed after radial sheath insertion and doppler ultrasound of the accesed radial artery was examined at the day after the procedure.

DETAILED DESCRIPTION:
Doppler ultrasound of the accessed artery was performed at the day after the radial procedure in all patients. The absence or presence of antegrade flow in the radial artery will be examined while compressing the ulnar artery as previously described.

The internal lumen radial artery diameter was evaluated by doppler ultrasound as the distance between the inner walls of the artery by personnel that are blinded to the study protocol.

Radial artery angiogram was performed soon after radial sheath insertion and the radial artery diameter was measured in AP projection in all patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing transradial catheterization

Exclusion Criteria:

* Systolic blood pressure < 100 mmHg

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2019-05-21 (Actual); Study Completion 2019-05-22 (Actual)

PRIMARY OUTCOMES:
The absence of antegrade radial artery flow by doppler evaluation | 24 hour
  The absence of radial artery flow by doppler evaluation
Blood pressure change | 2 minutes after drugs administration
  Blood pressure change after drugs administration

CONTACTS AND LOCATIONS:
Overall Officials: Surya Dharma, MD, PhD, Principal Investigator — Hermina Hospital Kemayoran
Locations (1):
- Hermina Heart Center, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dharma S, Kedev S, Patel T, Kiemeneij F, Gilchrist IC. A novel approach to reduce radial artery occlusion after transradial catheterization: postprocedural/prehemostasis intra-arterial nitroglycerin. Catheter Cardiovasc Interv. 2015 Apr;85(5):818-25. doi: 10.1002/ccd.25661. Epub 2014 Sep 13. PMID 25179153